CLINICAL TRIAL: NCT04018937
Title: Early HLA Matched Sibling Hematopoietic Stem Cell Transplantation for Children with Sickle Cell Disease: a Sickle Transplant Advocacy and Research Alliance (STAR) Trial
Brief Title: Early Human Leukocyte Antigen (HLA) Matched Sibling Hematopoietic Stem Cell Transplantation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Ann E. Haight, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00093513
Record Dates: First submitted 2019-07-10; First posted 2019-07-15 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Sickle Cell Disease
Keywords: Pediatrics; Hematopoietic stem cell transplantation; HLA matched sibling
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Alemtuzumab; fludarabine; fludarabine phosphate; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Reduced Intensity Conditioning with FAM (Experimental): Children with SCD will received reduced intensity conditioning with fludarabine, alemtuzumab and melphalan (FAM) during HSCT with a HLA matched sibling donor
  Interventions: Drug: Alemtuzumab; Drug: Fludarabine; Drug: Melphalan

INTERVENTIONS:
Drug: Alemtuzumab — Alemtuzumab will be administered by either subcutaneous (SQ) injection or IV. A test dose of alemtuzumab, 3 mg, is administered on the first day. If the test dose is tolerated, administration of three treatment doses will begin within 24 hours. The three treatment doses will be administered on consecutive days. On the first day, 10 mg/m2 will be given, 15 mg/m^2 the second and 20 mg/m^2 the third. Alemtuzumab will be started between Days -22 and -20, but all doses (test dose and three treatment doses) should be completed by Day -18.
  Other Names: Campath
Drug: Fludarabine — Fludarabine will be administered at 30 mg/m^2 IV daily for five days (Days -7 to -3).
  Other Names: Fludara
Drug: Melphalan — Melphalan will be administered at 140 mg/m^2 IV on Day -3 following fludarabine administration.
  Other Names: Alkeran; Evomela

SUMMARY:
This study aims to enroll 58 pre-adolescent (<13 years) pediatric participants with sickle cell disease (SCD) who have a pre-adolescent sibling bone marrow donor. All participants will go through a pre-transplant evaluation to find out if there are health problems that will keep them from being able to receive the transplant. It usually takes 2 to 3 months to complete the pre-transplant evaluation and make the arrangements for the transplant. Once they are found to be eligible for transplant, participants will be admitted to the hospital and will start transplant conditioning. Conditioning is the chemotherapy and other medicines given to prepare them to receive donor cells. It prevents the immune system from rejecting donor cells. Conditioning will start 21 days before transplant. Once they complete conditioning, participants will receive the bone marrow transplant. After the transplant, participants will stay in the hospital for 4-6 weeks. After they leave the hospital, participants will be followed closely in the clinic. Outpatient treatment and frequent clinic visits usually last 6 to 12 months. Routine medical care includes at least a yearly examination for many years after transplant by doctors and nurses familiar with sickle cell disease and transplant. The researchers will collect and study information about participants for 2 years after transplant.

DETAILED DESCRIPTION:
The use of HLA matched sibling donor (MSD) hematopoietic stem cell transplantation (HSCT) for sickle cell disease (SCD) is evolving. Because of the low risk for graft versus host disease (GVHD) associated with younger age, HSCT is increasingly being performed prior to adolescence. The use of less gonadotoxic reduced intensity regimens (RIC) are more commonly be utilized to lessen the risk for infertility. Finally, with the recognition that most children, even those who have asymptomatic to relatively mild courses, will develop debilitating morbidities as adults and ultimately suffer an early death, HSCT is being offered to children across a wider spectrum of SCD severity. Long reserved for severely affected children, HSCT is being performed for a growing number of less severely affected children, as well as children without disease manifestation.

This trial is designed to prospectively assess HSCT under these conditions. Eligibility will be limited to children less than 13 years of age who have an HLA MSD. A RIC regimen - fludarabine, alemtuzumab and melphalan (FAM) - will be employed. Finally, SCD severity criteria will be broadened to include less severely affected children as well as those who are severely affected.

This study has the following two specific aims:

Specific Aim #1: To prospectively assess the safety and efficacy of HSCT using FAM conditioning in children with SCD of varying severity who are under 13 years of age.

Specific Aim #2: To address current gaps in our understanding of the long-term effects of HSCT in children with SCD, by longitudinally assessing sickle cell related cerebrovascular disease, sickle cell related nephropathy and health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 2 years and less than 13 years old and have a sickle hemoglobinopathy.
* Patient must have an HLA identical sibling donor who is less than 13 years old. Sibling donors must not have any form of SCD. It is acceptable for the donor to carry a hemoglobinopathy trait.
* Patients must meet criteria for symptomatic SCD as defined below.

  * Severe disease:

    * Previous clinical stroke, defined as a neurological deficit lasting longer than 24 hours plus new finding on head CT or brain MRI/MRA.
    * Progressive silent cerebral infarction, as evidenced by serial MRI scans that demonstrate the development of a succession of lesions (at least two temporally discreet lesions, each measuring at least 3 mm in greatest dimension on the most recent brain MRI/MRA) or the enlargement of a single lesion, initially measuring at least 3 mm). Lesions must be visible on T2-weighted MRI sequences.
    * Abnormal TCD testing (confirmed elevated velocities in any single vessel of TAMMV > 200 cm/sec for non-imaging TCD)
    * Significant vasculopathy on MRA (greater than 50% stenosis of > 2 arterial segments or complete occlusion of any single arterial segment).
    * Frequent (at least 3 per year for preceding 2 years) painful vaso-occlusive episodes (defined as episode lasting at least 4 hours and requiring hospitalization or outpatient treatment with parenteral opioids). If patient is on hydroxyurea and its use has been associated with a decrease in the frequency of episodes, the frequency should be gauged from the 2 years prior to the start of hydroxyurea.
    * Recurrent (at least 3 in lifetime) acute chest syndrome events which have necessitated erythrocyte transfusion therapy.
    * Any combination of at least 3 acute chest syndrome episodes and vaso-occlusive pain episodes (defined as above) yearly for 3 years. If patient is on hydroxyurea and its use has been associated with a decrease in the frequency of episodes, the frequency should be gauged from the 3 years prior to the start of hydroxyurea.
  * Less severe disease: to qualify as having less severe disease, patients must not meet criteria for severe disease and must have one of the following:

    * Asymptomatic cerebrovascular disease, as evidenced by one the following: Silent cerebral infarction with at least one lesion measuring at least 3 mm in one dimension that is visible on two planes on the most recent brain MRI, or, cerebral arteriopathy, as evidenced by conditional TCD (TAMMV>170cm/sec but <200cm/sec) on two separate scans >2 weeks apart). If patient has a conditional TCD, then a brain MRI/MRA to evaluate for vasculopathy is required.
    * 2 or more painful vaso-occlusive episodes (in lifetime) requiring hospitalization or outpatient treatment with parenteral opioids.
    * 2 or more episodes of acute chest syndrome (in lifetime) irrespective of SCD modifying therapy administered.
    * Any combination of at least 3 acute chest syndrome episodes and vaso-occlusive pain episodes (defined as above, lifetime).
  * Patients with HbSS and HbSβ°thalassemia who have no clinical complications of their sickle cell disease and do not meet the criteria for less severe or severe disease.
* Participant's parent or legal guardian must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.
* Patient must have been evaluated and parent(s)/legal guardian, and the patient as age appropriate as determined by the treating center, adequately counseled regarding treatment options for SCD by a pediatric hematologist.
* Co-enrollment on STAR Project Sickle Cure (PSC) study is required for sites that are activated and participating in the study.

Exclusion Criteria:

* Bridging (portal to portal) fibrosis or cirrhosis of the liver.
* Parenchymal lung disease stemming from SCD or other process defined as a diffusing capacity of the lungs for carbon monoxide (DLCO; corrected for hemoglobin) or forced vital capacity of less than 45% of predicted. Children unable to perform pulmonary function testing will be excluded if they require daytime oxygen supplementation.
* Renal dysfunction with an estimated glomerular filtration rate (GFR) < 50% of predicted normal for age.
* Cardiac dysfunction with shortening fraction < 25%.
* Neurologic impairment other than hemiplegia, defined as full-scale intelligence quotient (IQ) of less than or equal to 70, quadriplegia or paraplegia, or inability to ambulate.
* Lansky functional performance score < 70%.
* Patient is HIV infected.
* Donor is HIV infected.
* Patient with unspecified chronic toxicity serious enough to detrimentally affect the patient's capacity to tolerate HSCT.
* Patient's parent(s) or legal guardian is unable to understand the nature and the risks inherent in the HSCT process.
* History of lack of adherence with medical care that would jeopardize transplant course.
* Donor who for psychological, physiologic, or medical reasons is unable to tolerate a bone marrow harvest or receive general anesthesia.
* Active viral, bacterial, fungal or protozoal infection.

  * Patients with viral upper respiratory tract infections should be asymptomatic for at least 7 days prior to enrollment. PCR testing for respiratory viruses (nasopharyngeal sample) should be negative at the start of the conditioning regimen. Exceptions may be made in patients with prolonged carriage (repeatedly positive over many weeks) of rhinovirus. These exceptions should be discussed with and approved by both study co-chairs and STAR Medical Director.

Ages: 2 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Immune Suppression-free, Rejection-free Survival | Year 2
  Immune suppression-free, rejection-free survival is defined as rejection-free survival off all systemic immunosuppressive agents. Participants who are off systemic immune suppression by 2-years post-transplant will be considered as being immune suppression free.

SECONDARY OUTCOMES:
Regimen-Related Toxicity | Day 42
  Regimen-Related Toxicity (RRT) will be scored according to the Bearman scale. Major RRT, defined as grade 4 (causing death) in any organ system or grade 3 for pulmonary, cardiac, renal, oral mucosal, neurologic or hepatic, will be recorded. The assessment for RRT will be carried out on day 42 post-transplant.
Number of Neurological Complications | Up to Year 2
  Neurological complications will be defined as any one of the following: seizures, intracranial hemorrhage, infarctive stroke (clinical or sub-clinical), and/or encephalopathy, including posterior reversible encephalopathy syndrome (PRES).
Neutrophil Recovery | Up to Year 2
  Neutrophil recovery is defined as the first of 3 consecutive days following the nadir that the absolute neutrophil count is at least 500/µl.
Platelet Recovery | Up to Year 2
  Platelet recovery is defined as the first day that the platelet count is at least 50,000/µl without a transfusion in the preceding 7 days.
Graft Rejection | Up to Year 2
  This endpoint will be met when donor engraftment fails to occur as evidenced by lack of neutrophil recovery or donor chimerism (5% donor derived cells on chimerism testing; for sorted testing, at least 5% of both lineages must be donor derived). This endpoint will also be met when there is initial donor engraftment but donor chimerism is lost.
Sustained Donor Engraftment | Year 2
  This endpoint will be met when the patient is off all immune suppression (or is still on immune suppression as treatment for GVHD) by one year, has normal marrow function, has no acute signs of SCD and has at least 5% donor derived cells on chimerism testing (for sorted testing at least 5% of both lineages must be donor derived). This endpoint will be assessed through 2 years.
Cytomegalovirus (CMV) Viremia | Day 180
  CMV Viremia will be defined as the occurrence of a positive polymerase chain reaction (PCR) test prior to day 180.
CMV Invasive Disease | Up to Year 2
  CMV invasive disease will be defined in accordance with the Blood and Marrow Transplant Clinical Trials Network Manual of Procedures.
Post-transplant Lymphoproliferative Disorder | Up to Year 2
  Post-transplant lymphoproliferative disorder will be defined in accordance with the Blood and Marrow Transplant Clinical Trials Network Manual of Procedures.
Other Infections | Up to Year 2
  Other Infections will be defined in accordance with the Blood and Marrow Transplant Clinical Trials Network Manual of Procedures.
Early Onset Acute GVHD | Day 100
  Early onset (before day 100) acute GVHD (including all grades, and stratified by grades) will be assessed according to the Blood and Marrow Transplant Clinical Trials Network Manual of Procedures using the NIH consensus criteria.
Late Onset Acute GVHD | Up to Year 2
  Late onset (after day 100) acute GVHD will be assessed according to the Blood and Marrow Transplant Clinical Trials Network Manual of Procedures using the NIH consensus criteria.
Chronic GVHD | Up to Year 2
  Chronic GVHD will be assessed according to the Blood and Marrow Transplant Clinical Trials Network Manual of Procedures using the NIH consensus criteria.
Rejection-free Survival | Up to Year 2
  Rejection-free survival is defined as survival with sustained engraftment.
Overall Survival | Up to Year 2
  Overall survival is defined as survival with or without rejection.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Haight, MD, Principal Investigator — Emory University
Locations (15):
- United States (13):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Children's, Phoenix, Arizona
  - Yale University, Yale Cancer Center, New Haven, Connecticut
  - Children's National Hospital, Washington D.C., District of Columbia
  - Children's Healthcare of Altanta, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Riley Children's Health/Indiana University, Indianapolis, Indiana
  - Dana-Farber Cancer Institute/Boston Children's Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Atrium Health Levine Cancer Institute, Charlotte, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Canada (2):
  - Cancercare Manitoba/Winnipeg Children's Hospital, Winnipeg, Manitoba
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leonard A, Furstenau D, Abraham A, Darbari DS, Nickel RS, Limerick E, Fitzhugh C, Hsieh M, Tisdale JF. Reduction in vaso-occlusive events following stem cell transplantation in patients with sickle cell disease. Blood Adv. 2023 Jan 24;7(2):227-234. doi: 10.1182/bloodadvances.2022008137. PMID 36240296